CLINICAL TRIAL: NCT06702306
Title: Duplex UltraSound afTer Endo Revascularisation - Feasibility Randomised Control Trial (DUSTER)
Acronym: DUSTER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other); Imperial College Healthcare NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 349192; RFPB207121 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2024-10-14; First posted 2024-11-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Limb Threatening Ischaemia
Keywords: Chronic limb threatening ischaemia; endovascular; ultrasound surveillance; randomised controlled trial
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Feasibility Randomised Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): At 1, 6 & 12 months post-procedure, patient will have specialist clinic appointment, with the following:
  * Wound inspection, pedal pulse palpation
  * Questionnaires to assess quality of life & pain (EQ5D-L, VASCUQOL-6, Barthel index, NRS-11)
- Ultrasound Surveillance Group (Experimental): Will receive the same care as control group, plus, lower limb arterial ultrasound, ankle and toe blood pressure checks before every in-person clinic appointment at 1, 6 & 12 months.
  Intervention arm participants are invited to take part in 1:1 interview with the research team after 6 months held as per participants' preference on MS Teams, via telephone, or in person.
  Interventions: Diagnostic Test: Ultrasound Surveillance

INTERVENTIONS:
Diagnostic Test: Ultrasound Surveillance — Lower limb arterial ultrasound, ankle and toe blood pressure checks before every in-person clinic appointment at 1, 6 and 12 months.
  Arms: Ultrasound Surveillance Group

SUMMARY:
17, 000 people every year in the UK develop foot pain or wounds from blocked leg arteries. If left untreated, this can lead to amputation. Keyhole surgery is often used to balloon open the blockages before they can cause serious problems. However half of people over the next 2 years can develop further blockages, which can be identified by ultrasound scans of the leg arteries

The aim of this clinical trial is to explore the benefits of regular ultrasound checks of the leg after keyhole surgery.

In this study participants are randomly allocated to one of two groups. Half of participants will have standard clinic appointments with their vascular specialist at 1 month, 6 months and 12 months. The other half will have additional ultrasound scans of the leg arteries before their clinic appointments at 1, 6 and 12 months.

We will then look at how many people attended the scans, whether the scans could be completed and how this affected decisions to have more surgery. At the end of the trial we will look at what happened to participants in both groups.

DETAILED DESCRIPTION:
Phase 1: Feasibility RCT

The study is a multi-site, randomised (1:1), controlled, open label, 2 arm, feasibility trial.

DUSTER will be performed in 3 NHS vascular units at the following NHS Trusts:

* Mid and South Essex NHS Foundation Trust
* Imperial College Healthcare NHS Trust
* Manchester University NHS Trust

These sites comprise two urban and one rural site, in both the North, South and East of the country. This will help understand the effects of travel, ethnicity, and geography on attending appointments. Following NIHR INCLUDE guidance we have costed for translation of study materials / interpreters.

Phase 2: Participant interviews

Participants in the intervention arm will be invited to individual semi-structured interviews with members of the research team. The interviews will be held as per participants' preference on MS Teams, or via telephone, or in person, after a minimum 6 month follow up.

The interviews seek to explore factors affecting adherence and the impact of integrated surveillance on patients. It will apply a Qualitative Descriptive Research (QDR) approach and aims to inquire into the experience of everyday living with chronic limb threatening ischaemia. QDR aims to provide broad insight into phenomena as experienced/lived by individuals and is widely used as the qualitative component in mixed-methodology studies especially in large-scale healthcare intervention studies to identify participants' perceptions of why ultrasound surveillance worked or did not work and how it might be better implemented. Using QDR in this manner can make modifications to how surveillance is delivered in a future HTA study, including behavioural modifications such as educational tools, automated reminders along with intervention modifications e.g. community-based scanning.

Phase 3: Participant and stakeholder focus groups

After the feasibility study, we will invite participants and stakeholders to 2 separate focus groups (face to face or MS teams-hybrid) to discuss potential secondary endpoints for a future HTA application (e.g. amputation free survival, quality of life and cost-effectiveness). These will be co-chaired with our lay co-applicants.

HTA application drafting

If progression criteria are met (see , Phases 1 -3 will feed into a draft HTA application in the final month of the study. The progression criteria are:

* >80% of ultrasound surveillance appointments are attended (>72/90), AND
* >90% completion rate of at least one ultrasound scan component (>81/90), AND
* There is an increase of >10% in re-interventions in ultrasound surveillance arm (>3 patients).

ELIGIBILITY:
Inclusion Criteria:

* Adults (18y+) who have had successful lower limb endovascular therapy (angioplasty, stenting, atherectomy, lithotripsy, drug eluting balloon or stent, or combination of above) for chronic limb threatening ischaemia (ischaemic rest pain, ulceration or gangrene with arterial imaging confirming peripheral arterial disease). Technical success is defined as <30% residual stenosis in the treated segments and patient leaving hospital without a major (above ankle) amputation on study leg
* Procedures within the last 3 weeks
* Interventions to iliac, femoral, tibial, and pedal vessels alone or in combination
* Endarterectomy or cutdown is permissible
* Able to give informed consent

Exclusion Criteria:

* Surgical bypass or endarterectomy alone undertaken
* Patient unfit for or does not want any future revascularisation
* Need for major amputation due to gas gangrene, severe Charcot deformity, extensive tissue loss with unstable foot, severe pedal disease on angiography or patient request
* Patient unwilling or cannot attend further surveillance
* Interventions for claudication or acute limb ischaemia or trauma
* Patients unable to take any form of antiplatelet therapy (aspirin or clopidogrel)
* Prior leg endovascular therapy at same anatomical location in study leg (within 1 year)
* Currently taking part in research that may impact on the results, design, or scientific value of this study or other studies that the potential participant may be taking part in.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess feasibility of ultrasound surveillance | 1 year
  * attendance at ultrasound surveillance appointments
  * completion rates of components of ultrasound surveillance
  * of participants undergoing arterial reintervention

SECONDARY OUTCOMES:
Limb Salvage | 1 year
  Limb salvage
Quality of Life | 1 Year
  Quality of Life measured via EQ5D-L questionnaire
Disease specific quality of life | 1 Year
  Disease specific quality of life measured via VASCUQOL-6 questionnaire
Independence in daily activities | 1 Year
  Independence in activities of daily living measured via the Barthel index
Participant reported pain | 1 Year
  Pain scores measured via NRS-11 questionnaire
Amputations | 1 Year
  Number and reasons for major amputation
Serious reintervention complications | 1 Year
  Serious reintervention complications (Clavien-Dindo Grade III-V)
Adverse events (cardiac/cerebrovascular) | 1 Year
  Major adverse cardiac or cerebrovascular events
Mortality | 1 Year
  Mortality and cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Ankur Thapar, PhD, Principal Investigator — Mid and South Essex NHS Foundation Trust
Locations (1):
- Mid & South Essex NHS Foundation Trust, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised outcome data for primary and secondary endpoints to 12 months will be made available for IPD meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: Ankur Thapar

REFERENCES:
- [Derived] Gadi N, Moore C, Hayden K, Zhang J, Beetar G, Rogers S, Smith-Ball C, Davies A, Thapar A. Duplex ultrasound after endo revascularisation (DUSTER): protocol for a randomised controlled feasibility trial. BMJ Open. 2025 Aug 10;15(8):e101137. doi: 10.1136/bmjopen-2025-101137. PMID 40784780